CLINICAL TRIAL: NCT04163419
Title: A Phase 2 Randomized, Double-blind, Placebo-Controlled Study of the Analgesic Efficacy and Safety of the Subcutaneous Administration of the Anti-NGF Antibody Tanezumab in Subjects With Moderate to Severe Pain Due to Schwannomatosis
Brief Title: Phase 2 Study of Tanezumab in Subjects With Moderate to Severe Pain Due to Schwannomatosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Scott R. Plotkin, MD, PhD, Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003201
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Schwannomatosis; Pain
Keywords: schwannoma; nerve growth factor; antibody; NGF
MeSH Terms: conditions — Schwannomatosis; Pain; Neurilemmoma; Hereditary Sensory and Autonomic Neuropathies | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (treatment) (Experimental): Tanezumab 10 mg SC administered on day 1 and Day 57 (± 4 days)
  Interventions: Drug: Tanezumab
- Arm B (placebo then treatment) (Placebo Comparator): Placebo SC (to match tanezumab SC) administered on Day 1 and tanezumab 10 mg SC on Day 57 (± 4 days)
  Interventions: Drug: Tanezumab; Drug: Placebo

INTERVENTIONS:
Drug: Tanezumab — Tanezumab 10 mg SC
  Other Names: PF-04383119
Drug: Placebo — Placebo 10 mg SC
  Arms: Arm B (placebo then treatment)

SUMMARY:
The primary objective of this study is to determine whether the administration of tanezumab, an anti-nerve growth factor (NGF) antibody, improves pain relief in schwannomatosis patients receiving background non-NSAID therapy.

DETAILED DESCRIPTION:
Schwannomatosis is characterized by the predisposition to develop multiple schwannomas and, less commonly, meningiomas. Pain is the most frequent symptom reported by these patients, with 68% experiencing chronic pain.

The investigators propose to test the efficacy and tolerability of tanezumab as a treatment for schwannomatosis patients with chronic pain who have had inadequate pain relief in a randomized, placebo-controlled trial, which could form the basis of a larger, randomized controlled trial in the future.

The study is designed with a total duration of 281 days (40 weeks) and will consist of four periods: Pre-treatment, Double-Blind Treatment, Single Arm Treatment, and 24-Week Safety Follow-up. The Pre-Treatment Period lasting up to 30 days, followed by a Double-Blind Treatment Period lasting up to 8 weeks, followed by a Single Arm Treatment Period lasting up to 8 weeks, and a 24-Week Safety Follow-Up Period ending with the End of Study Visit at Week 40.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis schwannomatosis by fulfilling either clinical or molecular diagnosis.
2. Age ≥ 18 years. Patients < 18 years are excluded since the safety profile of tanezumab in this population has not been determined.
3. ECOG performance status ≤2 or Karnofsky ≥60%
4. Participants must have normal organ and marrow function as defined per the full protocol
5. The subject's weight must be≥ 45 kg at Screening.
6. The subject must be willing to avoid prohibited pain medications (including non-steroidal anti-inflammatory drugs) throughout the duration of the study except as permitted per Protocol.
7. Subject must have moderate to severe pain secondary to schwannomatosis, defined as Score ≥5 on the Numeric Rating Scale-11 (NRS-11) at Screening.
8. Subject must have failure, intolerance, or contraindication to at least three standard of care therapies:

   * Documented history indicating that NSAID therapy has not provided adequate pain relief or subject is unable to take NSAIDs due to contraindication or inability to tolerate.
   * Documented history indicating that opioid treatment has not provided adequate pain relief or subject is unwilling to take opioids, or unable to take opioids due to contraindication or inability to tolerate
   * Documented history indicating that neuropathic pain medications, such as gabapentin, pregabalin, or others, have not provided adequate pain relief or subject is unable to take these treatments due to contraindication or inability to tolerate.
9. Female subjects of childbearing potential and at risk for pregnancy (e.g., not abstinent) must agree to use 2 highly effective methods of contraception throughout the study and for 112 days (16 weeks) after the last dose of assigned subcutaneous study medication.

Exclusion Criteria:

1. Subjects with any of the following criteria: evidence of bilateral vestibular schwannomas on imaging, a known germline pathogenic NF2 mutation, a first-degree relative who meets diagnostic criteria for NF2, or have schwannomas limited to a previous radiation field.
2. Subjects with intracranial meningioma associated with cerebral edema on neuroimaging. Note: presence of intracranial meningioma itself is not an exclusion criterion.
3. Subjects who have had surgery, chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) for treatment of a painful schwannomatosis-related tumor prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
4. Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days (or 90 days for biologics) before Screening and/or during study participation.
5. Subjects receiving anticoagulation to treat an underlying medical condition.
6. Subject has a history of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG fusion protein.
7. The subject's pain is related to a non-schwannomatosis cause such as prior cancer therapy, infection, bowel obstruction/perforation, spinal cord compression, or fracture or impending fracture of weight bearing bone.
8. The subject has a diagnosis of malignancy in the last 3 years (except for Gleason 6 prostate cancer, basal cell carcinoma or carcinoma in situ).
9. Use of concurrent adjuvant analgesics such as serotonin norepinephrine reuptake inhibitors (SNRI), tricyclic antidepressants, anticonvulsant medication, or muscle relaxants (unless the drugs were started at least 30 days prior to Screening and are maintained at a stable dose).
10. Use of concurrent analgesic non-steroidal anti-inflammatory drugs (NSAIDs, including selective COX-2 inhibitors) unless the subject is expected to be able to discontinue these medications at least 2 weeks prior to treatment. Note: Subjects who take daily low dose aspirin (≤ 325 mg as per local prescribing practice) therapy for cardiovascular prophylaxis are not excluded from participation.
11. Diagnosis of osteoarthritis of the knee or hip as defined by the American College of Rheumatology (ACR) combined clinical and radiographic criteria; Radiographic criteria will be assessed by the Central Reader.
12. Use of concurrent corticosteroids (except for inhaled or topical corticosteroids as needed for management of ongoing pulmonary or dermatologic conditions)
13. Subjects considered unfit for surgery, defined as Grade >3 on the American Society of Anesthesiologists (ASA) physical classification system for surgery or subjects who would not be willing to undergo joint replacement surgery if required.
14. Subjects with symptoms and radiographic findings (i.e. joint space narrowing, osteophytes) consistent with osteoarthritis in the shoulder.
15. History of significant trauma or surgery to a major joint (e.g. hip, knee or shoulder) within one year prior to Screening.
16. A history of osteonecrosis or osteoporotic fracture (i.e., a subject with a history of osteoporosis and a minimally traumatic or atraumatic fracture).
17. Radiographic (x-ray) evidence of any of the following conditions as determined by the central radiology reviewer at Screening: 1) rapidly progressive osteoarthritis, 2) atrophic or hypotrophic osteoarthritis, 3) subchondral insufficiency fracture, 4) spontaneous osteonecrosis of the knee (SPONK), 5) osteonecrosis, or 6) pathologic fracture.
18. Subjects who have evidence of orthostatic hypotension based upon replicate orthostatic blood pressure measurements at Screening.
19. Subjects with a total impact score of >7 on the Survey of Autonomic Symptoms (SAS) at Screening.
20. Diagnosis of a transient ischemic attack in the 6 months prior to Screening or diagnosis of stroke with residual deficits (e.g., aphasia, substantial motor or sensory deficits), that would preclude completion of required study activities.
21. History, diagnosis, or signs and symptoms of clinically significant neurological
22. Subjects with a past history of carpal tunnel syndrome (CTS) with signs or symptoms of CTS in the one year prior to Screening.
23. Subject with a history of significant alcohol, analgesic, or narcotic substance abuse within the six months prior to Screening.
24. Subject who, in the judgement of the investigator, is expected to require a surgical procedure during the duration of the study.
25. Previous exposure to exogenous nerve growth factor or to an anti-nerve growth factor antibody.
26. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the trial
27. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
28. Pregnant females; breastfeeding females; females of childbearing potential not using two (2) methods of highly effective contraception or not agreeing to continue two (2) methods of highly effective contraception for 112 days (16 weeks) after last dose of investigational product.
29. Any subject who, in the judgement of the investigator, is deemed inappropriate for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain level | 8 weeks
  Change in worst pain level during past week from baseline to week 8 measured by NRS-11

SECONDARY OUTCOMES:
Frequency of AEs | 40 weeks
  Frequency of AEs related to treatment with Tanezumab
Incidence of orthostatic hypotension | 40 weeks
  Incidence of orthostatic hypotension using postural changes in blood pressure in addition to mean changes in postural blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Plotkin, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Da JLW, Merker VL, Jordan JT, Ly KI, Muzikansky A, Parsons M, Wolters PL, Xu L, Styren S, Brown MT, Plotkin SR. Design of a randomized, placebo-controlled, phase 2 study evaluating the safety and efficacy of tanezumab for treatment of schwannomatosis-related pain. Contemp Clin Trials. 2022 Oct;121:106900. doi: 10.1016/j.cct.2022.106900. Epub 2022 Aug 26. PMID 36038003